CLINICAL TRIAL: NCT02057861
Title: The Comparison of Reversal of Neuromuscular Blockade in Diabetic and Non-Diabetic Patients
Brief Title: Reversal of Neuromuscular Blockade in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, yavuz demiraran, Professor Doctor, Duzce University
Other Study IDs: ozlemersoy
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Observation of Neuromuscular Block
Keywords: diabetes mellitus; neuromuscular blockade; sugammadex
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non-diabetic: non-diabetic group; 2 mg/kg sugammadex iv, postoperatively Extubation times were recorded.
- diabetic: Diabetic group; 2 mg/kg sugammadex iv, postoperatively Extubation times were recorded

SUMMARY:
In this study the investigators aimed to compare the time of antagonism and intensity of effect of sugammadex which is used for antagonism of rocuronium on diabetic and non-diabetic patients.

DETAILED DESCRIPTION:
Aim: In this study the investigators aimed to compare the time of antagonism and intensity of effect of sugammadex which is used for antagonism of rocuronium on diabetic and non-diabetic patients.

Methods: Included patients were divided into 2 groups: diabetic (n=21) and non-diabetic (n=20). All patients were premedicated. After arrival in the operating room, all patients were monitorised with Datex Ohmeda S/5 Anesthesia Machine and electrocardiography (DII derivation), hemodynamic variables, respiratory rate, and inspiratory sevoflurane concentrations were recorded. Neuromuscular monitoring system was used. Anesthesia was induced with propofol 2 mg/kg and fentanyl 1 mcg/kg. After the loss of eyelid reflex the neuromuscular monitoring system automatically identified supramaximal stimulating currents and after that rocuronium 0,6 mg/kg was given. Train of four (TOF) stimulation with the supramaximal current were applied and by recording of second TOF value (TOF2) the patient was intubated. Anesthesia was maintained with 50% O2 + 50% air and sevoflurane of 1-2 % concentration. TOF stimulation was applied and recorded every 20 seconds. Intraoperatively by return T2 rocuronium 0,15 mg/kg was given. T2i time was recorded as intubation time and T2d time was recorded as clinical effect time. At the end of the operation sugammadex 2 mg/kg was given. When TOF rate reached 0,9 patients were extubated and the time was recorded.

ELIGIBILITY:
Inclusion Criteria:

* The patients (diabetic and non-diabetic) between 18-65 years with risk of anesthesia I-II,
* For diabetic group patients with Diabetes mellitus Type 2 over 10 years.
* For non-diabetic group patients without any glucose metabolism disease

Exclusion Criteria:

* myasthenia gravis, myotonic dystrophia, motor neuron diseases
* diabetic neuropathy and nephropathy
* hepatic, renal and cardiac diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients (diabetic and non-diabetic) between 18-65 years
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
reversal of diabetic patients | 24 hours
  T2i time was recorded as intubation time and T2d time was recorded as clinical effect time. At the end of the operation sugammadex 2 mg/kg was given. When TOF rate reached 0,9 patients were extubated and the time was recorded.

SECONDARY OUTCOMES:
hemodynamic changes | 24 hours
  Systolic, diastolic blood pressure and heart rate were recorded in the peroperative period

CONTACTS AND LOCATIONS:
Overall Officials: yavuz demiraran, professor, Principal Investigator — Duzce University
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)